CLINICAL TRIAL: NCT06733402
Title: A Multi-center, Double-blind, Randomized, Placebo Controlled, Parallel-group Study, Comparing Trifarotene Cream 0.005% (Taro Pharmaceuticals U.S.A, Inc.) to Aklief® Cream (US REFERENCE LISTED DRUG), Aklief Cream (REFERENCE PRODUCT) and Each Active Treatment to a Placebo Control in the Treatment of Acne Vulgaris.
Brief Title: A Study Comparing Trifarotene Cream 0.005% to AKLIEF® CREAM (US REFERENCE LISTED DRUG), AKLIEF™ CREAM (CANADIAN REFERENCE PRODUCT) in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRFC-2405
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Trifarotene Cream 0.005% (Experimental): A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Interventions: Drug: Trifarotene Cream 0.005%
- AKLIEF® Cream (Trifarotene 0.005%) US REFERENCE LISTED DRUG (Active Comparator): A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Interventions: Drug: AKLIEF® Cream (Trifarotene 0.005%) US REFERENCE LISTED DRUG
- AKLIEF® Cream (Trifarotene 50 mcg/g) CANADIAN REFERENCE PRODUCT (Active Comparator): A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Interventions: Drug: AKLIEF® Cream (Trifarotene 50 mcg/g) CANADIAN REFERENCE PRODUCT
- Placebo Control (Placebo Comparator): A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trifarotene Cream 0.005% — A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Other Names: Test Product
  Arms: Trifarotene Cream 0.005%
Drug: AKLIEF® Cream (Trifarotene 0.005%) US REFERENCE LISTED DRUG — A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Other Names: Reference Product
  Arms: AKLIEF® Cream (Trifarotene 0.005%) US REFERENCE LISTED DRUG
Drug: AKLIEF® Cream (Trifarotene 50 mcg/g) CANADIAN REFERENCE PRODUCT — A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Other Names: Reference Product
  Arms: AKLIEF® Cream (Trifarotene 50 mcg/g) CANADIAN REFERENCE PRODUCT
Drug: Placebo — A thin layer of the investigational product will be self-applied to the affected areas of the face once daily at bedtime.
  Other Names: Vehicle
  Arms: Placebo Control

SUMMARY:
To demonstrate the efficacy, therapeutic equivalence and safety of Trifarotene Cream 0.005% (Taro Pharmaceuticals U.S.A., Inc.) and US Reference Listed Drug, Canadian Reference Product over the placebo control in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, placebo-controlled, parallel-group study, comparing comparing Trifarotene Cream 0.005% (Taro Pharmaceuticals U.S.A, Inc.) to Aklief® Cream (US REFERENCE LISTED DRUG), Aklief Cream (REFERENCE PRODUCT) and each active treatment to a placebo control in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Subjects must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3 or 4 as per the Investigator's Global Assessment (IGA).
* Subjects must have ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 20 inflammatory lesions (i.e., papules and pustules) AND ≤2 nodulocystic lesions (i.e., nodules and cysts), at baseline on the face.
* Subjects must be willing to refrain from using all other topical acne medications or antibiotics for acne vulgaris during the 12-week treatment period, other than the investigational product.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Subjects with a history of hypersensitivity or allergy to Trifarotene, retinoids and/or any of the study medication ingredients.
* Subjects with excessive facial hair (e.g. beards, sideburns, mustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris.
* Subjects with a baseline irritation score of 3 = severe (marked, intense).

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Demonstrate the therapeutic equivalence, efficacy and safety of the Investigational Product | Baseline to Week 12
  Percentage change in the inflammatory (papules and pustules) & non-inflammatory (open and closed comedones) of the lesion counts.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals, Inc.
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No